CLINICAL TRIAL: NCT03042325
Title: Prospective, Multi-center, Open-label, Phase IV Study to Evaluate the Safety and Efficacy of Alogliptin as Monotherapy or Add on Therapy in Indian Patients With Type 2 Diabetes Mellitus
Brief Title: Safety and Efficacy of Alogliptin in Indian Participants With Type 2 Diabetes Mellitus
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Business decision, no safety or efficacy concerns
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SYR-322-4001; U1111-1174-1852 (Registry Identifier: WHO)
Record Dates: First submitted 2017-02-01; First posted 2017-02-03 (Estimated); Last update posted 2017-10-20 (Actual); Status verified 2017-10

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Drug therapy
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — alogliptin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Alogliptin (Experimental): Alogliptin 25 mg, tablets, orally, once, daily for 26 weeks in addition to standard care for the management of Type 2 Diabetes Mellitus (T2DM). Dose will be adjusted as per creatinine clearance [CrCl].
  Interventions: Drug: Alogliptin

INTERVENTIONS:
Drug: Alogliptin — Alogliptin tablets
  Other Names: SYR-322; Nesina

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of alogliptin tablets when given as monotherapy or add on therapy in participants who are on standard care for management of Type 2 Diabetes Mellitus (T2DM).

DETAILED DESCRIPTION:
The drug being tested in this study is called alogliptin. Alogliptin is being tested to treat people who have Type 2 Diabetes Mellitus (T2DM). This study will look at side effects and glycemic control in people who take alogliptin in addition to standard care.

The study will enroll approximately 300 patients. All participants will receive alogliptin tablets at a dose determined based on the creatinine clearance.

The recommended dose of alogliptin is 25 mg once daily with normal or mildly impaired renal function (creatinine clearance [CrCl] ≥60 mL/min), dose of 12.5 mg for participants with moderate renal impairment (CrCl ≥30 to <60 mL/min), and 6.25 mg for participants severe renal impairment (CrCl ≥15 to <30 mL/min). Participants with end-stage renal disease (ESRD) (CrCl <15 mL/min or requiring hemodialysis) will be excluded, in addition to standard care for the management of T2DM.

All participants will be asked to take one tablet every morning each day throughout the study.

This multi-center trial will be conducted in India. The overall time to participate in this study is up to 33 weeks. Participants will make multiple visits to the clinic, and will be contacted by telephone 30 days after last dose of study drug for a follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Participants with T2DM who are dipeptidyl peptidase-4 (DPP-4) inhibitor-naive; including alogliptin.

Exclusion Criteria:

1. Has contraindication or limitation for administration of alogliptin tablets according to the approved label/Prescribing Information.
2. Participants treated with alogliptin tablets outside the approved label/ prescribing information.
3. Has end-stage renal disease (ESRD) (Creatinine Clearance (CrCl) <15 mL/min or requiring hemodialysis).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-07-30 (Estimated); Primary Completion 2018-01-15 (Estimated); Study Completion 2018-01-15 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants with Adverse Events (AEs) and Serious Adverse Events (SAEs) | Baseline up to 30 days after the last dose of study drug (up to 30 weeks)
  An Adverse Event (AE) is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (example, a clinically significant abnormal laboratory finding), symptom, or disease temporally associated with the use of a drug, whether or not it is considered related to the drug. A serious adverse event (SAE) is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; or congenital anomaly; or a medically important event.
Percentage of Participants with Adverse Drug Reactions (ADRs) and Unexpected ADRs | Baseline up to 30 days after the last dose of study drug (up to 30 weeks)
  An ADR is any response to a medicinal product which is noxious and unintended and which occurs at doses normally used in man for the prophylaxis, diagnosis or therapy of diseases or for the restoration, correction or modification of physiological function. Response in this context means that a causal relationship between a medicinal product and an adverse event is at least a reasonable possibility.
Change from Baseline in Glycosylated Haemoglobin (HbA1c) at Weeks 13 and 26 | Baseline and Weeks 13 and 26
  The change in the value of glycosylated hemoglobin (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound) collected at weeks 13 and 26 relative to Baseline.
Percentage of Participants with Glycosylated Hemoglobin < 7.0% | Weeks 13 and 26
  Clinical response at Weeks 13 and 26 will be assessed by the percentage of participants with HbA1c less than 7%.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director Clinical Science, Study Director — Takeda